CLINICAL TRIAL: NCT05233761
Title: Le Rêve 3.0: A Double-Blind, Placebo-Controlled, Randomized, Crossover Investigational Study to Determine if Defined CBD, a Capsule With a Custom Formulation of Cannabidiol (CBD) and Terpenes, Influences Sleep Physiology
Brief Title: Evaluation of an Oral Cannabidiol (CBD)-Terpene Formulation on Sleep Physiology in Participants With Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Defined Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DR-INS-101
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: Cannabidiol
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Defined CBD (Experimental): Defined CBD will be administered as two small capsules that will be taken orally with a glass of water one hour before bedtime that contain a total of 300 mg CBD and 8 mg terpenes. Participants will take the treatment on a minimum of four nights per week, over a total of four-weeks.
  Interventions: Drug: Defined CBD
- Placebo (Placebo Comparator): The placebo control will be administered as two small capsules that will be taken orally with a glass of water one hour before bedtime that do not contain any CBD or terpenes. Participants will take the treatment on a minimum of four nights per week, over a total of four-weeks. The Placebo capsules will look and smell identical to the Defined CBD capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Defined CBD — 300 mg CBD and 8 mg Terpenes administered as two small capsules.
  Arms: Defined CBD
Drug: Placebo — Capsules that smell and look exactly like Defined CBD but contain no CBD or terpenes.
  Arms: Placebo

SUMMARY:
Insomnia is a disorder in which people have inadequate or poor-quality sleep due to a number of factors, such as difficulty falling asleep, waking up frequently during the night with difficulty returning to sleep, waking up too early in the morning, or having unrefreshing sleep. Defined CBD is a capsule composed of highly purified (>99.9%) hemp-derived cannabidiol (CBD) and terpenes produced as a potential sleep aid for people with insomnia. This product contains no detectable Delta-9-tetrahydrocannabinol (Delta-9-THC). This trial is specifically designed to evaluate the efficacy of Defined CBD on sleep physiology in people with insomnia.

DETAILED DESCRIPTION:
Our research study aims to test the effects of a highly purified CBD product on the structure and function of sleep physiology. In a survey by Consumer Reports, ~40% of adults who reported trying CBD said they used it to help them sleep, and a majority of those people said it worked. Nonetheless, to this date a rigorous, properly-controlled, and well-powered study to determine if CBD influences sleep physiology has simply never been reported in the scientific literature. The Le Rêve 3.0 study is designed to fill this important void in scientific knowledge.

We hypothesize that a novel CBD-based formulation in the form of an orally administered capsule will positively impact sleep physiology in subjects with insomnia. The capsule we will test is composed of >99.9% purity hemp-derived CBD with a custom chemical formulation that also contains low concentrations (1 mg each) of highly purified (>98%) forms of the terpenes linalool, myrcene, phytol, limonene, alpha-terpinene, alpha-terpineol, alpha-pinene, and beta-caryophyllene. Preclinical studies in animals have shown that these terpenes are sedating, but their potential effects on sleep physiology in humans have not been established. This product contains no detectable Delta-9-THC.

The Le Rêve 3.0 study will involve a cross-over design in which study participants will cycle through two independent treatments each for four weeks (Treatment 1: Placebo; Treatment 2: Defined CBD). The study participants will initially be randomized with respect to the treatment group, and all participants will be cycled through each of the two treatments. We will use a double-blind design in which the investigator and study participants will both be blinded to the treatments. Baseline data for each participant will be collected for two weeks prior to initiating treatments, as well as for a one-week washout period following each treatment arm. The entire study will last 12 weeks.

The primary objective of the study is to determine if Defined CBD influences objective measures of sleep physiology. Primary sleep physiology data will be obtained in a completely unbiased manner from a non-invasive sleep-tracking wristband, called "Whoop" (https://www.whoop.com), that electronically collects and transmits sleep data from study participants in the comfort of their own beds. The wristband collects hundreds of data points per second from a 3-axis accelerometer, 3-axis gyroscope, and heart rate sensor. The wristband can accurately measure latency to fall asleep, total sleep time, sleep fragmentation, as well as the time spent in each sleep stage [Light, Slow Wave (Deep), Rapid Eye Movement (REM), and Awake]. The wristband also collects data using photoplethysmography (PPG), a technique that involves measuring blood flow by assessing superficial changes in blood volume. Heart rate, heart rate variability, and respiratory rate, can all be derived from PPG data, and all of these metrics are used in Whoop's sleep detection and staging algorithms. Importantly, two recent publications, published independently from Whoop, show that data on sleep stages collected from the Whoop device are highly accurate and correlate well with polysomnography (PSG), the gold-standard of sleep tracking used in clinical studies conducted in sleep clinics.

The secondary objective of the study is to determine if Defined CBD influences subjective measures of sleep physiology. We will collect this subjective data from study participants in the form of a brief five-minute survey that will be completed on their smartphone at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided a signed and dated informed consent form.
2. Presence of chronic insomnia defined as self-reported difficulty initiating (latency to persistent sleep >30 min) and/or maintaining sleep (>30 mins awake during the middle of the night, or waking >30 mins before desired waking time on three or more nights per week) for at least 3 months.
3. Insomnia Severity Index score >15.
4. Male or female aged 25-70 years.
5. Is willing to comply with all study procedures throughout the entire study, including:

   * Wearing a sleep-tracking device on their wrist throughout entire clinical study.
   * Ensuring that the sleep-tracking device is connected to their smartphone via Bluetooth on a daily basis so that sleep data can be collected on a daily basis.
   * Ensuring that the sleep-tracking device is charged before going to bed each night, ensuring that sleep data can be collected on a daily basis.
   * Is willing to receive and respond to daily text (SMS) notifications for the duration of the entire clinical study.
   * During the treatment phases of the study, is willing to take the treatment for at least four nights in each week.
6. On the nights in which the participant takes the treatment, is willing to abstain from excessive alcohol intake (>two drinks/day).
7. On the nights in which the participant takes the treatment, is willing to refrain from drinking alcohol two hours before bedtime.
8. Female subjects who:

   * Are postmenopausal, with amenorrhea for at least one year before the screening interview, OR
   * Are surgically sterile, OR
   * If of childbearing potential agree to practice effective double barrier methods of contraception (e.g., condom + diaphragm; condom or diaphragm + spermicidal gel or foam), from the time of the signing of informed consent through the last dose of study treatment, or agree to completely abstain from intercourse.
9. Self-reported bedtime between 9 pm and midnight on four-seven nights per week.
10. Owns a smartphone.

Exclusion Criteria:

1. Self-reported body mass index > 32 calculated from patient's height (m) and weight (kg); weight (kg)/square height (m²).
2. Insomnia associated with clinically diagnosed sleep apnea (AHI greater than 15 events/hour), or movement disorders such as restless legs, periodic limb movement (PLM) (greater than 30 events/hour or greater than five events/hour with associated PLM arousals).
3. Are currently participating in a formal behavioral therapy program to facilitate sleep.
4. History of epilepsy or seizures.
5. History of liver disease.
6. Serious head injury or stroke within the past year.
7. Psychiatric disorders including major depression, bipolar, anxiety, or schizophrenia.
8. History of suicide attempt or current suicide ideation.
9. Evidence of any clinically significant, severe or unstable, acute or chronically progressive medical or surgical disorder (including planned medical procedures that may impact sleep), or any condition that may interfere with the absorption, metabolism, distribution, or excretion of the study drug.
10. Patients with a history of cardiovascular disease including poorly controlled hypertension, ischemic heart disease, arrhythmia, or severe heart failure.
11. Untreated metabolic disorder such as diabetes.
12. Medical conditions that result in frequent need to get out of bed (e.g. nocturia).
13. History of drug or alcohol abuse, including past or present history of cannabis dependence.
14. Inability to refrain from greater than two standard drinks/day of alcohol consumption for study duration.
15. Current cigarette smoker.
16. Currently chronic (daily) cannabis user.
17. Use of any substance with psychotropic effects or properties known to affect sleep/wake, including neuroleptics, morphine/opioid derivatives, antihistamines, stimulants, anti-depressants, clonidine, within one week prior to screening.
18. Use of any over-the-counter sleep medications including tryptophan, valerian root (Valeriana officinalis), kava (Piper methysticum Forst), melatonin, St John's Wort (Hypericum perforatum), Alluna (herbal sleep supplement with valerian root), and hemp within one week prior to screening.
19. Inability to refrain from use of any of the following contra-indicated drugs for at least one week prior to and for the duration of the study: erythromycin, clarithromycin, itraconazole, ketoconazole, posaconazole, voriconazole, ritonavir, telaprevir, boceprevir, amlodipine, gemfibrozil, cyclosporine, danazol, amiodarone, verapamil, diltiazem, rifampin, theophylline, tizanidine, bupropion, efavirenz, diflunisal, propofol, fenofibrate, lamotrigine, morphine, lorazepam, diazepam, clobazam, stiripentol, valproate, everolimus, sirolimus, or tacrolimus, niacin (vitamin B3 greater than 1g/ day), grapefruit juice.
20. Consumption of xanthine-containing beverages (i.e., tea, coffee, energy drinks or cola) of more than five cups or glasses per day.
21. Inability to refrain from greater than 400mg/day of caffeine consumption for study duration.
22. Participation in any other clinical trial within 30 days before the screening visit.
23. Night shift workers (during the 12 months prior to the study and during the study).
24. Individuals who nap three or more times per week over the preceding month.
25. Current delayed sleep phase syndrome where wake-up time is regularly (>5x/week) later than 9:00 a.m.
26. Individuals having to travel across more than two time zones or outside of their country of residence at any time during the study.
27. Females who are pregnant, are planning to become pregnant, or are breastfeeding.
28. History of allergies particularly to plant-based products containing terpenes, i.e. flavors and aromatic natural oils for example citrus, mango, lavender, thyme, cedarwood and pine products.
29. Known hypersensitivity to cannabinoids, including CBD.
30. Individuals may be excluded from participating in the study based on the investigator's professional judgement.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 125 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Muchowski, Ph.D., Principal Investigator — Defined Research Institute
Locations (1):
- Defined Research, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang M, Faust M, Abbott S, Patel V, Chang E, Clark JI, Stella N, Muchowski PJ. Effects of a cannabidiol/terpene formulation on sleep in individuals with insomnia: a double-blind, placebo-controlled, randomized, crossover study. J Clin Sleep Med. 2025 Jan 1;21(1):69-80. doi: 10.5664/jcsm.11324. PMID 39167421

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (A to B: A = Placebo; B = Defined CBD): The placebo control will be administered as two small capsules that will be taken orally with a glass of water one hour before bedtime that do not contain any CBD or terpenes. Participants will take the treatment on a minimum of four nights per week, over a total of four-weeks. The Placebo capsules look and smell identical to the Defined CBD capsules.
  Defined CBD will be administered as two small capsules that will be taken orally with a glass of water one hour before bedtime that contain 300 mg CBD and 8 mg terpenes. Participants will take the treatment on a minimum of four nights per week, over a total of four-weeks.
- Group 2 (B to A: B = Defined CBD; A = Placebo): Defined CBD will be administered as two small capsules that will be taken orally with a glass of water one hour before bedtime that contain 300 mg CBD and 8 mg terpenes. Participants will take the treatment on a minimum of four nights per week, over a total of four-weeks.
  The placebo control will be administered as two small capsules that will be taken orally with a glass of water one hour before bedtime that do not contain any CBD or terpenes. Participants will take the treatment on a minimum of four nights per week, over a total of four-weeks. The Placebo capsules look and smell identical to the Defined CBD capsules.
Period: Treatment Period A
Arm/Group | Group 1 (A to B: A = Placebo; B = Defined CBD) | Group 2 (B to A: B = Defined CBD; A = Placebo)
Started | 63 | 62
Completed | 37 | 25
Not Completed | 26 | 37
Not completed — Withdrawal by Subject | 12 | 10
Not completed — Lost to Follow-up | 6 | 12
Not completed — Protocol Violation | 8 | 15
Period: Treatment Period B
Arm/Group | Group 1 (A to B: A = Placebo; B = Defined CBD) | Group 2 (B to A: B = Defined CBD; A = Placebo)
Started | 37 | 25
Completed | 37 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (A to B: A = Placebo; B = Defined CBD) | Group 2 (B to A: B = Defined CBD; A = Placebo) | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 62 | 125
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 50 | 101
  Male | 12 | 12 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent in the Combination of Slow Wave Sleep (SWS) and Rapid Eye Movement (REM) Sleep
Description: The primary endpoint is the percentage of time spent in slow wave (Deep) and REM sleep as quantified by a non-invasive wrist-worn sleep-tracking device called Whoop.
Time Frame: Participants were assessed for treatment with CBD-terpenes and placebo, each for a treatment period of four weeks. Participants took the treatment (CBD-terpenes or Placebo) for at least four nights per week over the entire four week treatment period.
Population: Data from six participants [four participants from Group 1 (A/B) and two participants from Group 2 (B/A)] were excluded from the final data analysis due to protocol deviations (e.g. due to a lack of reporting whether or not they took the study treatment, and/or insufficient sleep data collection).
Measure: Mean (Standard Error); unit: Percentage of total sleep time
Arm/Group | Defined CBD | Placebo
Number analyzed (Participants) | 56 | 56
Percentage of total sleep time | 43.0 (0.4) | 41.8 (0.4)
Statistical Analysis 1: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in SWS + REM (% TST) sleep in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in SWS + REM sleep (% TST) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority; p = 0.0350, t-test, 2 sided; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.1 to 2.5], Standard Error of Mean 0.6

2. Secondary Outcome: Objective Secondary Outcome Measures of Sleep Physiology
Description: The percentage of time spent in each sleep stage (SWS, REM, light and awake) relative to total sleep time as quantified by a non-invasive wrist-worn sleep-tracking device called Whoop.
Time Frame: Four weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage of TST
Arm/Group | Defined CBD | Placebo
Number analyzed (Participants) | 56 | 56
Percentage of TST
  SWS Sleep (%TST) | 19.1 (0.2) | 18.1 (0.2)
  REM Sleep (% TST) | 24.0 (0.3) | 23.7 (0.3)
  Light Sleep (% TST) | 56.0 (0.4) | 57.7 (0.4)
  Awake Time (% TST) | 22.4 (0.5) | 21.7 (0.4)
Statistical Analysis 1: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in SWS Sleep (% TST) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in SWS Sleep (% TST) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.0019, t-test, 2 sided; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.4 to 1.6], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in REM Sleep (% TST) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in REM Sleep (% TST) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.52, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-.6 to 1.2], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in Light Sleep (% TST) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in Light Sleep (% TST) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.0040, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.8 to -0.5], Standard Error of Mean 0.6
Statistical Analysis 4: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in Awake Time (% TST) sleep in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in Awake Time (% TST) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.24, t-test, 2 sided; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-.5 to 2.0], Standard Error of Mean 0.6

3. Secondary Outcome: Objective Secondary Outcome Measures of Sleep Physiology
Description: The absolute time spent in each sleep stage (SWS, REM, light and awake) as quantified by a non-invasive wrist-worn sleep-tracking device called Whoop.
Time Frame: Four weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Min
Groups:
- Defined CBD: Defined CBD will be administered as two small capsules that will be taken orally with a glass of water one hour before bedtime that contain 300 mg CBD and 8 mg terpenes. Participants will take the treatment on a minimum of four nights per week, over a total of four-weeks.
Arm/Group | Defined CBD | Placebo
Number analyzed (Participants) | 56 | 56
Min
  SWS+REM Sleep (min) | 162.5 (2.0) | 155.0 (2.2)
  SWS Sleep (min) | 71.1 (0.9) | 67.7 (1.0)
  REM Sleep (min) | 91.4 (1.4) | 90.0 (1.5)
  Light Sleep (min) | 206.2 (2.5) | 212.9 (2.6)
  Awake Time (min) | 80.4 (1.7) | 78.2 (1.7)
  Total Sleep Time (min) | 366.5 (3.3) | 373.4 (3.3)
Statistical Analysis 1: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in SWS + REM Sleep (min) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in SWS + REM Sleep (min) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.0117, t-test, 2 sided; Mean Difference (Final Values) = 4.9, 95% CI 2-sided [1.7 to 13.3], Standard Error of Mean 2.6
Statistical Analysis 2: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in SWS Sleep (min) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in SWS Sleep (min) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.0126, t-test, 2 sided; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [0.7 to 5.9], Standard Error of Mean 1.3
Statistical Analysis 3: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in REM Sleep (min) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in REM sleep (min) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.51, t-test, 2 sided; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.7 to 5.3], Standard Error of Mean 2.0
Statistical Analysis 4: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in Light Sleep (min) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in Light Sleep (min) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.0574, t-test, 2 sided; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-13.7 to 0.2], Standard Error of Mean 3.6
Statistical Analysis 5: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in Awake Time (min) in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in Awake Time (min) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.3, t-test, 2 sided; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-2.4 to 6.9], Standard Error of Mean 2.4
Statistical Analysis 6: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in Total Sleep Time (min) sleep in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in Total Sleep Time (min) in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment difference in percentages was estimated and constructed using the above-mentioned method; p = 0.14, t-test, 2 sided; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-16.1 to 2.4], Standard Error of Mean 4.7

4. Secondary Outcome: Subjective Secondary Outcome Measure of Sleep Physiology
Description: A modified version of a clinically validated questionnaire/survey entitled the patient's global impression (PGI) was used to assess subjective perceptions of sleep by the study participants after each four-week treatment period. The modified PGI is a five-item, subjective, participant self-report that assesses treatment benefit to sleep quality (Item 1), sleep induction (Item 2), sleep duration (Item 3), sleep depth (Item 4) and treatment effect on the presence of vivid dreams (item 5). Each item in our modified PGI was presented as a survey that consisted of a ten-point categorical scale, with scores between 6-10 representing a treatment benefit/advantage, a score of 5 representing no effect of treatment, and a score of 1-4 representing a treatment worsening/disadvantage.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Defined CBD | Placebo
Number analyzed (Participants) | 56 | 56
Units on a scale
  Sleep Better | 5.9 (0.4) | 5.6 (0.4)
  Sleep Induction | 5.6 (0.4) | 5.1 (0.4)
  Sleep Duration | 5.6 (0.4) | 4.8 (0.4)
  Sleep Depth | 5.5 (0.4) | 5.0 (0.4)
  Vivid Dreams | 4.5 (0.5) | 4.0 (0.5)
Statistical Analysis 1: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in the perception of "better sleep" in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in the perception of "better sleep" in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment differences was estimated and constructed using the above-mentioned method; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-.7 to 1.3], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in the perception of "sleep induction" in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in the perception of "sleep induction" in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment differences was estimated and constructed using the above-mentioned method; p = 0.32, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.6 to 1.7], Standard Error of Mean 0.6
Statistical Analysis 3: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in the perception of "sleep duration" in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in the perception of "sleep duration" in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment differences was estimated and constructed using the above-mentioned method; p = 0.20, t-test, 2 sided; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.4 to 1.9], Standard Error of Mean 0.6
Statistical Analysis 4: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in the perception of "sleep depth" in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in the perception of "sleep depth" in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment differences was estimated and constructed using the above-mentioned method; p = 0.45, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.7 to 1.6], Standard Error of Mean 0.6
Statistical Analysis 5: Comparison: Defined CBD vs Placebo; The null hypothesis was that there was no difference in the perception of "vivid dreams" in participants that received CBD-terpenes and the placebo control; the alternative hypothesis was that there was a significant difference among the two treatment groups; Test type: Superiority — The mean nightly difference in the perception of "vivid dreams" in participants that received CBD-terpenes and the placebo control at the end of the two four-week treatment phases was analyzed using a two-sided test with an alpha level at 0.05 to evaluate superiority. The P-value and 95% confidence interval for the estimate of treatment differences was estimated and constructed using the above-mentioned method; p = 0.4, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.8 to 1.9], Standard Error of Mean 0.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected on a daily basis by a medical monitor throughout the 12 week duration of the study.
Description: The definitions of adverse events and/or serious adverse events that were used to collect adverse event information were identical to those described by clinical trials.gov.
Arm/Group | Defined CBD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/88
Other Adverse Events (participants affected / at risk) | 0/99 | 0/88

LIMITATIONS AND CAVEATS:
First, the study was not conducted in a sleep clinic using polysomnography. Second, the wrist-worn sleep-tracking device used in the current study does not measure sleep latency and may not be sufficiently accurate to report sleep staging. Third, the unexpected high dropout rate in the study limited its statistical power, especially with respect to subjective outcome measures of sleep.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT05233761/Prot_SAP_001.pdf